CLINICAL TRIAL: NCT06711081
Title: Clinical and Radiographic Evaluation Following Complete Pulpotomy Using Low Level LASER Therapy and Cryotherapy
Brief Title: Clinical & Radiographic Efficacy Using LLLT & CRYO on M.P.M Pulpotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mohamed motiea mohamed morsy, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLLT& CRYO pulpotomy on M.P.M
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: MTA Vital Tooth Pulpotomy
Keywords: vital pulp therapy permanent teeth pulpotomy LLLT
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group I: Conventional complete Pulpotomy using MTA (control group). (No Intervention): MTA putty material will be placed using premixed capsule which will be triturated according to manufacturer's instructions. MTA will be placed in a 2-3 mm layer above the pulp tissue using an amalgam carrier and gently packed to the canal orifice using a condenser, then it will be covered by moistened cotton pellet for 2 minutes to achieve the initial setting, then the cotton pellet will be removed. A layer of resin modified glass ionomer cement will be placed and the tooth will be restored using light cured composite filling material .
- • Group II: LLLT following complete pulpotomy. (Active Comparator): after achieving homeostasis, LLLT will be applied using diode laser of 810 nm wave length with energy of 2 J/cm2 under a continuous mode with power output of 100 mW for about 10 sec with laser tip size 600 μm and 2 mm away from the canal orifice, Then MTA will be placed and the tooth will be restored as in group I.
  Interventions: Device: low level laser device cryotherapy
- • Group III: Cryotherapy following complete pulpotomy. (Active Comparator): after achievement of homeostasis, the cryotherapy will be applied using small piece of shaved sterile ice wrapped with sterile piece of gauze (0° Celsius) which will be placed over the pulpal tissue in the pulp chamber. After approximately 60 seconds, the molten ice will be removed, then MTA will be placed and the tooth will be restored as in group I.
  Interventions: Device: low level laser device cryotherapy

INTERVENTIONS:
Device: low level laser device cryotherapy — using new device direct on the pulp tissue
  Other Names: cryotherapy
  Arms: • Group II: LLLT following complete pulpotomy.; • Group III: Cryotherapy following complete pulpotomy.

SUMMARY:
This in-vivo study aims to evaluate the efficacy of the low level laser therapy and cryotherapy in treatment of vital pulpotomy in mature permanent molar evaluating the post operative pain and the radiographic changes in pulpal and periodontal regions.

DETAILED DESCRIPTION:
Recently, there is a new direction of vital pulp therapy (VPT) that aims to preserve the tooth vitality and the root dentin and improves the long term prognosis of the tooth function. VPT is a personalized method of treating irreversible pulpitis which conforms to the trend of minimally invasive endodontics. There are many modalities of VPT like direct pulp capping, indirect pulp capping, pulpotomy and revascularization. Pulpotomy is defined as clinical procedure of removal of the coronal pulp tissue leaving the vital radicular pulp tissue as in cases of pulp exposure due to caries, trauma or iatrogenic error. Pulpotomy may be complete or partial according to the degree of extension of pulpal inflammation.

VPT depends on the theory that the pulp has the capacity of self-healing when it is free from infection. In addition, recent innovations of dental materials and techniques have been administrated to the field of endodontics have ensured higher success rate of VPT. Pulpotomy procedure has been introduced as an alternative to traditional root canal treatment in case of mature permanent teeth exhibiting symptoms of irreversible pulpitis when the radicular pulp is still vital.

There are many materials and techniques used for pulpotomy where the selection of the material used for this technique greatly influences its success rate. An ideal material for VPT must be biocompatible, antibacterial, providing biological and bacterial tight seal and promoting the regeneration of dentine-pulp complex. Calcium hydroxide (Ca(OH)2) and mineral trioxide aggregate (MTA) are considered the most commonly used materials for pulpotomy. However, Ca(OH)2 has many drawbacks as degradation over time, formation of tunnel defects beneath dentinal bridges and poor sealing ability, so it has lost its popularity as a first choice agent for pulpotomy. On the other hand, MTA has better sealing ability, biocompatibility and strength. However, it has some drawbacks like difficult handling, long setting time and discoloration of the tooth.

More recent pulpotomy materials have been introduced as putty bioceramic materials including: calcium silicate, monobasic calcium phosphate, zirconium oxide, tantalum oxide, and filler agents. They show better handling due to its premixed putty consistency in addition to its low level of tooth discoloration and rapid setting time compared to MTA.

In addition to the new materials, there are modifications of pulpotomy techniques which has been administrated to enhance its outcome as light amplification of estimated emission of radiation (LASER) and cryotherapy. The application of laser may enhance the outcomes of pulpotomy due to its ability to vaporize water in dental hard tissue so dentinal tubules will be opened and smear layer will be removed which in turn will increase the sealing ability of pulpotomy material.

One of the special forms of laser application is called low level laser therapy (LLLT) which can act as photoactivator on the pulp tissue cells by photostimulation without heat formation to enhance the cell differentiation and dentinogensis stimulation to promote tissue healing. In addition, it shows comparable effect to non-steroidal anti-inflammatory drugs (NASIDS), so it can be considered as an alternative to pain control through reduction of the exudative phase of inflammatory process, increasing synthesis of endorphins, decreasing bradykinin and altering pain threshold. On the other hand, the main disadvantages of laser include its uncontrolled depth of penetration through the tissue in addition to high cost of the laser device.

Moreover, Cryotherapy is another modified technique for pulpotomy. It is a procedure used to destroy tissue by freezing or re-thawing process through decreasing the temperature of the tissue. It has several physiological responses as decreasing of the local blood flow which can affect the homeostasis, temporary inhibition of the neural receptors in the pulp and decreasing of metabolic activity which in turn may affect the post-operative pain.

Cone beam computed tomography (CBCT) can be used for determination of periapical-periodontal status as it provides three dimensional demonstrations of the anatomic features plus accurate dimensional readings of the periapical tissue. The success of pulpotomy can be evaluated through the periapical-periodontal status radiographically which is confirmed clinically by absence of signs and symptoms.

Post-operative pain after pulpotomy is common. It is a noxious feeling after doing the procedure which may start immediately or later. Effective management of the post-operative pain is important in reducing the recovery time and improving patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* • Restorable vital and mature mandibular molar teeth with irreversible pulpitis.

  * Teeth with deep caries or large restoration.
  * Pre-operative radiograph showing normal periapical structure.
  * Teeth with normal periodontal status .

Exclusion Criteria:

* • Medically compromised patients with active systemic disease as uncontrolled diabetes mellitus, hypertension or cardiac diseases.

  * Teeth with periapical lesion.
  * Sinus tract or swelling.
  * Moderate or severe marginal periodontitis.
  * Patient allergic to any material or medication used in this study.
  * Teeth with moderate to severe mobility.
  * Teeth with periodontal diseases.
  * Teeth with anatomical variations.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
radiographic changes | one year after treatment
  and x-ray change either pulpal or periapical using CBCT subtraction

SECONDARY OUTCOMES:
Post operative pain | one week after treatment
  Post operative pain using visual analog scale by the patient description pain on his own words

CONTACTS AND LOCATIONS:
Overall Officials: abeer darrag, phd, Principal Investigator — Professor of Endodontics; tokka moukhatar, Study Director — Lecturer of Endodontics
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray PE. Review of guidance for the selection of regenerative endodontics, apexogenesis, apexification, pulpotomy, and other endodontic treatments for immature permanent teeth. Int Endod J. 2023 Mar;56 Suppl 2:188-199. doi: 10.1111/iej.13809. Epub 2022 Aug 15. PMID 35929348
- [Background] Duncan HF, El-Karim I, Dummer PMH, Whitworth J, Nagendrababu V. Factors that influence the outcome of pulpotomy in permanent teeth. Int Endod J. 2023 Mar;56 Suppl 2:62-81. doi: 10.1111/iej.13866. Epub 2022 Nov 22. PMID 36334098